CLINICAL TRIAL: NCT01855269
Title: A Prospective Randomized Controlled Study: Lactobacillus Reuteri Versus Herbal Drop in the Treatment of Infantile Colic
Brief Title: Lactobacillus Reuteri Versus Herbal Drop in the Treatment of Infantile Colic: a Prospective Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Sami Ulus Children's Hospital (Other)
Responsible Party: Principal Investigator, Dilek Dilli, Assoc Prof, Dr. Sami Ulus Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 134/Feb 2012
Record Dates: First submitted 2013-05-13; First posted 2013-05-16 (Estimated); Last update posted 2013-05-16 (Estimated); Status verified 2013-05

CONDITIONS: Crying
Keywords: probiotic; infantile colic
MeSH Terms: conditions — Crying; Colic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lactobacillus reuteri (Active Comparator): Lactobacillus reuteri (BioGaia, Stockholm, Sweden):at a dose of 100 million colony forming unit in 5 drops, 30 minutes after feeding, once per day for 3 weeks
  Interventions: Dietary Supplement: Lactobacillus reuteri
- Herbal drop (Active Comparator): Herbal drop containing sodium bicarbonate, Pimpinella anisum oil, foeniculum vulgare oil, Mentha piperita (Babs, Berko, Istanbul, Turkey):5 drops 30 minutes after feeding, once per day for 3 weeks
  Interventions: Dietary Supplement: Herbal drop
- Sterile water (Placebo Comparator): Sterile water: 5 drops, 30 minutes after feeding, once per day for 3 weeks
  Interventions: Dietary Supplement: placebo sterile water

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri — Lactobacillus reuteri (BioGaia, Stockholm, Sweden):at a dose of 100 million colony forming unit in 5 drops, 30 minutes after feeding, once per day for 3 weeks
  Other Names: Biogaia
  Arms: Lactobacillus reuteri
Dietary Supplement: Herbal drop — Herbal drop containing sodium bicarbonate, Pimpinella anisum oil,foeniculum vulgare oil, Mentha piperita (Babs, Berko, Istanbul, Turkey):5 drops 30 minutes after feeding, once per day for 3 weeks
  Other Names: Babs
  Arms: Herbal drop
Dietary Supplement: placebo sterile water
  Arms: Sterile water

SUMMARY:
The aim was to test the hypothesis that oral administration of Lactobacillus reuteri in a prospective randomized controlled study would improve symptoms of infantile colic.

DETAILED DESCRIPTION:
Infantile colic ıs one of the most common problems within the first 3 months of life, affecting as many as 3% to 28% of newborn children. It consists of a behavioral syndrome characterized by paroxysmal, excessive, inconsolable crying without identifiable cause. Lactobacillus reuteri, one of the few endogenous lactobacillus species in the human gastrointestinal tract, has been used safely for many years as a probiotic dietary supplement in adults, and recent data demonstrated safety after long-term dietary supplementation for newborn infants. The positive effects of this probiotic on intestinal disorders such as constipation and diarrhea and in protection from infection,as well as its capacity to modulate immune responses.

The aim was to test the hypothesis that oral administration of Lactobacillus reuteri in a prospective randomized controlled study would improve symptoms of infantile colic.

ELIGIBILITY:
Inclusion Criteria:

* infants three weeks to three months
* infants with colic three hours of crying on three days in the week
* infants feeding with breast milk
* infants weighing 2500 to 4000 gram

Exclusion Criteria:

* chronic illness
* gastrointestinal disorders
* infants received either antibiotics or probiotics in the previous week

Ages: 3 Weeks to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 74 (Actual)
Dates: Start 2012-04; Primary Completion 2013-02 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Crying time | 3 weeks
  Infants crying episodes, feeding and stooling characteristics, growth, weight gain were noted weekly for three weeks

SECONDARY OUTCOMES:
postpartum depression | 3 weeks
  Emotional structures of mother's behaviour were evaluated before and at 2nd month with Edinburgh postpartum depression scale (EPDS), State Trait Anxiety Inventory (STAI) tests.

CONTACTS AND LOCATIONS:
Overall Officials: Nilgün Karadağ, MD, Principal Investigator — MD, Sami Ulus CH
Locations (1):
- Sami Ulus CH, Ankara, Turkey, Turkey (Türkiye)

REFERENCES:
- [Result] Savino F, Pelle E, Palumeri E, Oggero R, Miniero R. Lactobacillus reuteri (American Type Culture Collection Strain 55730) versus simethicone in the treatment of infantile colic: a prospective randomized study. Pediatrics. 2007 Jan;119(1):e124-30. doi: 10.1542/peds.2006-1222. PMID 17200238